CLINICAL TRIAL: NCT01847131
Title: Effectiveness of Oxymetazoline Added on Intranasal Steroid in the Treatment of Allergic and Nonallergic Rhinitis With Persistent Nasal Obstruction
Brief Title: Effectiveness of Oxymetazoline Added on Nasal Steroid in Rhinitis With Persistent Nasal Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R015532021
Record Dates: First submitted 2013-04-14; First posted 2013-05-06 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Nasal Obstruction Present Finding
Keywords: Rhinitis; Oxymetazoline
MeSH Terms: conditions — Nasal Obstruction; Rhinitis | interventions — Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxymetazoline (Active Comparator): 0.05% oxymetazoline nasal sprays 2 sprays in each nostril twice daily
  Interventions: Drug: oxymetazoline
- placebo (Placebo Comparator): placebo nasal spray 2 sprays in each nostril twice daily
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: oxymetazoline — 0.05% Oxymetazoline nasal sprays were commercially available.
  Other Names: Iliadin
  Arms: oxymetazoline
Drug: Placebo nasal spray — Placebo nasal spray has made by the local pharmaceutical company in thailand who commercially manufacture and sell 0.05% oxymetazoline nasal spray. The placebo contains the same ingredients as the drug except the active ingredient.
  Arms: placebo

SUMMARY:
Background Allergic rhinitis is a common health problem with a worldwide prevalence is 10-25%, and poses significant impact on the quality of life of the patients. In Thailand, the prevalence of allergic rhinitis in the general population is 13.5%, of which the frequency of allergic rhinitis increased from 23% to 38% in the children, and 61.9% in the graduate students. Despite intranasal steroid being the current first-line treatment of patients with allergic rhinitis, only 60% of patients achieve excellent control. Persistent nasal congestion is the major symptom which is difficult to control in these patients. Data are limited about efficacy and safety of the additional use of 0.05% intranasal oxymetazoline hydrochloride (OXY) for persistent nasal congestion that does not adequately respond to recommended doses of intranasal steroid (INS) and oral antihistamine(OAH).

Objective To determine the efficacy and safety of the additional use of OXY for persistent nasal congestion in allergic rhinitis or non-allergic rhinitis patients inadequately controlled by combination treatment with INS and OAH.

Methods The investigators performed a 6-week, randomized, double blind, placebo controlled, clinical trial in 50 patients with allergic rhinitis or non-allergic rhinitis whom inadequately controlled by combination treatment with INS and oral antihistamine (OAH). After an initial screening, qualified individuals were randomized into 2 groups including the treatment group and the control group. The treatment group received the INS (2 puffs in each nostril twice daily) and OAH (1 tablet once daily) plus OXY (2 puffs in each nostril twice daily) The control group received INS (2 puffs in each nostril twice daily) and OAH (1 tablet once daily) plus placebo (2 puffs in each nostril twice daily).

DETAILED DESCRIPTION:
All participants will continue medications for 4 weeks, then stop using interventional medication and still take INS (2 puffs in each nostril twice daily) and OAH (1 tablet once daily) for 2 more weeks. Then, all participants will come for the last visit to see whether rebound nasal symptoms occur. Participants will be asked to record nasal symptom diary card, and nasal peak inspiratory flow. Rhinoconjunctivitis Quality of life Questionnaire (Rcq) will be recorded during visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or greater
* Diagnosis with allergic or nonallergic rhinitis with persistent nasal obstruction
* Being treated with intranasal steroid and oral antihistamine

Exclusion Criteria:

* Underlying disease of hypertension
* Use oral or nasal decongestant 7 days prior to entering the study
* Nasal polyp or significant deviated nasal septum
* Respiratory tract infection 14 days prior to entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torpong Thongngarm, M.D., Principal Investigator — Mahidol University; Panitan Pradubpongsa, M.D., Study Chair — Mahidol University; Paraya Assanasen, M.D., Study Chair — Mahidol University; Pongsakorn Tantilipikorn, M.D., Study Chair — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients from medical clinic were instructed to record the severity of nasal congestion 3 days prior to randomization. The severity of nasal congestion was recorded on a 0 to 3 scale (0 = no symptom and 3 = severe symptom). Participants who had nasal congestion score of 1 or greater were recruited for randomization.
Pre-assignment Details: Exclusion if patients with a history suggestive of cardiovascular, hepatic or renal diseases, pregnant or lactating women, taking oral or nasal decongestant within 7 days, treated with immunotherapy, patients with nasal polyp or significant deviated nasal septum and patient with a history of upper respiratory tract infection within 14 days.
Period: Overall Study
Arm/Group | Oxymetazoline | Placebo
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis were performed to compared between 2 groups on age, gender results of allergy skin tests and baseline nasal congestion scores.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxymetazoline | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants] — Age, gender, allergy skin prick testing for aeroallergens and baseline nasal congestion scores were measured.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 24 | 24 | 48
    >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Thailand | 25 | 25 | 50
nasal congestion scores [Geometric Mean (Standard Deviation); unit: units on a scale] — The severity of nasal congestion was recorded on a 0 to 3 scale (0 = no symptom, 1= mild symptom, 2 = moderate symptom and 3 = severe symptom).
  units on a scale | 1.73 (0.54) | 1.78 (0.64) | 1.76 (0.59)

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Oxymetazoline in the Treatment of Rhinitis With Persistent Nasal Obstruction
Description: Primary outcome measure is the nasal congestion score measuring by visual analog scale (VAS) ranging from 1-10 (0 = no symptom and 10 = the most severe symptom) compared between treatment group and controlled group.
Time Frame: 6 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oxymetazoline | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | 1.38 [0.95 to 1.81] | 1.67 [1.19 to 2.15]

2. Secondary Outcome: The Numbers of Subjects Who Developed Rhinitis Medicamentosa After Using Oxymetazoline
Description: Rhinitis medicamentosa is the rebound nasal congestion after prolonged use (>7 days) of topical nasal decongestant (eg. oxymetazoline). However, a previous study by Baroody FM et al (J Allergy Clin Immunol 2011;127:927-34) showed that using oxymetazoline together with intranasal steroid for 1 month did not increase rhinitis medicamentosa compared to placebo. So we give rhinitis patients in the treatment group with oxymetazoline and intranasal steroid for 1 month, then stop using oxymetazoline and come back for the last visit 2 weeks later to see which patients develop rebound nasal congestion (rhinitis medicamentosa).
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Oxymetazoline | Placebo
Number analyzed (Participants) | 25 | 25
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Oxymetazoline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 17/25 | 20/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxymetazoline (N=25) | Placebo (N=25)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9) — Upper respiratory tract infection including common cold, pharyngitis, etc
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) — Nasal discomfort includes nasal irritation and nasal pain.
Headache (Nervous system disorders) | 1 (1) | 3 (3) — Headache includes functional headache without localizing signs.
Insomnia (General disorders) | 1 (1) | 0 (0) — Difficulty of sleep without other specific symptoms.
Numbness at lips or tongue (General disorders) | 1 (1) | 1 (1) — The sense of numbness at lips or tongue without neurological localizing sign.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Epistaxis due to local irritation.

LIMITATIONS AND CAVEATS:
Further studies with larger numbers of subjects and longer period of follow-up would probably have led to significant differences between both treatment groups in NPIF, Rcq scores and the possible rebound nasal congestion or other adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No